CLINICAL TRIAL: NCT04133168
Title: Safety and Effectiveness IDE Trial for Boston Scientific's Cryoballoon in the Treatment of Symptomatic Drug Refractory Paroxysmal Atrial Fibrillation
Brief Title: Boston Scientific's Cryoballoon in the Treatment of Symptomatic Drug Refractory Paroxysmal Atrial Fibrillation
Acronym: FROZEN-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PY004
Record Dates: First submitted 2019-10-03; First posted 2019-10-21 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: cryoablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: open label, prospective, single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Cryoablation (Experimental): Subjects undergoing cardiac ablation procedure with the Boston Scientific Cardiac Cryoablation System
  Interventions: Device: Boston Scientific Cardiac Cryoablation System

INTERVENTIONS:
Device: Boston Scientific Cardiac Cryoablation System — The Boston Scientific Cardiac Cryoablation System is intended for ablation and electrical mapping of the pulmonary veins for pulmonary vein isolation (PVI) in the ablation treatment of patients with paroxysmal atrial fibrillation (PAF).The main devices and components of the system consists of the following:
  * POLARx™ or POLARx™ FIT Cryoablation Catheter
  * POLARMAP™ Catheter
  * POLARSHEATH™
  * SMARTFREEZE™ Console
  * Diaphragm Movement Sensor (DMS)
  * Related Accessories

SUMMARY:
To establish the safety and effectiveness of the Boston Scientific Cardiac Cryoablation System for treatment of symptomatic, drug refractory, recurrent, paroxysmal atrial fibrillation (AF).

DETAILED DESCRIPTION:
Multi-center, open label, prospective, single arm study to document the safety and performance of Boston Scientific's Cryoablation System. The Cryoablation System is intended for cryoablation and electrical mapping of the pulmonary veins for pulmonary vein isolation (PVI) in the ablation treatment of patients with paroxysmal atrial fibrillation (PAF). All subjects fitting the enrollment criteria, signing the consent and undergoing the index procedure with the study devices will be followed up for twelve (12) months after the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* History of recurrent symptomatic paroxysmal atrial fibrillation (PAF), defined as atrial fibrillation that terminates spontaneously or with intervention (either procedure or drug therapy) within seven days of onset. Minimum documentation includes the following:

  * a physician's note indicating recurrent self-terminating atrial fibrillation (AF) which includes at least two symptomatic AF episodes within six months prior to enrollment, and one electrocardiographically documented AF episode within 12 months prior to enrollment.
* No amiodarone use within 90 days prior to enrollment;
* Subjects who are indicated for an ablation procedure for paroxysmal atrial fibrillation (PAF) according to 2017 HRS expert consensus statement on catheter and surgical ablation of atrial fibrillation;
* Subjects refractory or intolerant to at least one class I or III antiarrhythmic medication;
* Subjects who are willing and capable of providing informed consent;
* Subjects who are willing and capable of participating in all testing associated with this clinical investigation at an approved clinical investigational center;
* Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* Any known contraindication to an AF ablation or anticoagulation;
* Continuous AF lasting longer than seven (7) days from onset;
* History of previous left atrial ablation or surgical treatment for AF/ AFL/ AT;
* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause;
* Structural heart disease or implanted devices as described below:

  1. Left ventricular ejection fraction (LVEF) < 40% based on the most recent transthoracic echocardiogram (TTE) (≤180 days prior to enrollment);
  2. Left atrial diameter > 55 mm OR left atrial volume > 50 ml/m2 ml indexed based on the most recent TTE (≤ 180 days prior to enrollment);
  3. An implanted pacemaker, ICD, CRT device or an arrhythmia loop recorder;
  4. Previous cardiac surgery: i.e. ventriculotomy or atriotomy (excluding atriotomy for CABG);
  5. Previous cardiac valvular surgical or percutaneous procedure, or prosthetic valve, including mitral valve clips;
  6. Interatrial baffle, closure device, patch, or patent foramen ovale (PFO) occlude;
  7. Presence of a left atrial appendage occlusion device;
  8. Presence of any pulmonary vein stents;
  9. Coronary artery bypass graft (CABG), PTCA/ PCI/ coronary stent procedures within 90 days prior to enrollment;
  10. Unstable angina or ongoing myocardial ischemia;
  11. myocardial infarction within 90 days prior to enrollment;
  12. Moderate or severe mitral insufficiency assessed on the most recent TTE (≤180 days prior to enrollment, e.g. pulmonary artery pressure >30 mmHg);
  13. Evidence of left atrial thrombus;
* Any previous history of cryoglobulinemia;
* Stage 3B or higher renal disease (estimated glomerular filtration rate, eGFR <45 mL/min);
* History of blood clotting or bleeding disease;
* Any prior history of documented cerebral infarct, TIA or systemic embolism [excluding a post-operative deep vein thrombosis (DVT)] ≤180 days prior to enrollment;
* Active systemic infection;
* Pregnant, lactating (current or anticipated during study follow up), or women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion);
* Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the sponsor to determine eligibility;
* Subjects who in the judgment of the investigator have a life expectancy of less than two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ellenbogen, MD, Study Chair — VCU Pauley Heart Center, Richmond, Virginia, USA; Arash Aryana, MD, PhD, Principal Investigator — Mercy General Hospital,Sacramento, CA , USA; Nassir Marrouche, MD, Principal Investigator — University of Utah School of Medicine. Slat Lake City, UT, USA; Ante Anić, MD, Principal Investigator — University Hospital, Split, Croatia; Suneet Mittal, MD,FACC,FHRS, Principal Investigator — Snyder AF Center, New York, NY, USA; Niraj Varma, MD,PhD,FRCP, Principal Investigator — Cleveland Clinic, Cleveland OH, USA; Wilber W Su, MD,FACC,FHRS, Principal Investigator — Banner- University Medical Group- Heart Center, Phoenix, AZ, USA
Locations (44):
- United States (30):
  - Banner University Medical Center, Phoenix, Arizona
  - Pima Heart and Vascular, Tucson, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Cedars - Sinai Medical Center, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - Torrance Memorial Medical Center, Torrance, California
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - AdventHealth Tampa, Tampa, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Southcoast Physicians Group, Fall River, Massachusetts
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Valley Hospital, Ridgewood, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Northwell Health, Staten Island, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Stern Cardiovascular Foundation, Inc., Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - Chippenham & Johnston-Willis Hospital, Richmond, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - PeaceHealth Southwest Medical, Vancouver, Washington
  - St. Mary's Medical Center, Huntington, West Virginia
  - Aurora Health Care, Grafton, Wisconsin
- UZ Brussels, Brussels, Belgium
- Canada (4):
  - Hamilton General Hospital, Hamilton, Ontario
  - Institut de Cardiologie de Montreal, Montreal
  - Institut universitaire de Cardiologie et de Pneumologie de Quebec, Québec
  - Vancouver General Hospital, Vancouver
- CHU Grenoble - Hopital Michallon, Grenoble, France
- Germany (2):
  - Herz-und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Maria Cecilia Hospital SPA, Cotignola, Italy
- Erasmus MC- University Medical Center Rotterdam, Rotterdam, Netherlands
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei, Beitou District
  - National Taiwan University Hospital, Taipei, Zhongzheng Dist

IPD SHARING:
Plan to Share IPD: No
No requests for study data have been made at this time, however Boston's Scientific's policy on data sharing can be found at http://www.bostonscientific.com/en-US/data-sharing-requests.html

REFERENCES:
- [Result] Ellenbogen KA, Mittal S, Varma N, Aryana A, Marrouche N, Anic A, Nair D, Champagne J, Iacopino S, de Asmundis C, Weiner S, Makati K, Raybuck JD, Richards E, Su W. One-year outcomes of pulmonary vein isolation with a novel cryoballoon: Primary results of the FROZEN AF trial. J Cardiovasc Electrophysiol. 2024 Apr;35(4):832-842. doi: 10.1111/jce.16220. Epub 2024 Mar 6. PMID 38448797

RESULTS

PARTICIPANT FLOW:
Groups:
- FROzEN: Subjects undergoing cardiac ablation procedure with the Boston Scientific Cardiac Cryoablation System
  Boston Scientific Cardiac Cryoablation System: The Boston Scientific Cardiac Cryoablation System is intended for ablation and electrical mapping of the pulmonary veins for pulmonary vein isolation (PVI) in the ablation treatment of patients with paroxysmal atrial fibrillation (PAF).The main devices and components of the system consists of the following:
  * POLARx™ or POLARx FIT Cryoablation Catheter
  * POLARMAP™ Catheter
  * POLARSHEATH™
  * SMARTFREEZE™ Console
  * Diaphragm Movement Sensor (DMS)
  * Related Accessories
Period: FROzEN AF Clinical Study
Arm/Group | FROzEN
Started | 404 (63 Roll-In subjects; 336 Non Roll-In subjects; 5 consent ineligible)
Procedure | 326 (Treatment = 325; Attempt = 1)
Pre-Discharge | 325
7 Day Follow Up | 321 (Missed =3)
3 Month Follow Up | 315 (Missed=6)
6 Month Follow Up | 310 (Missed = 9)
12 Month Follow Up | 308
Completed | 308
Not Completed | 96
Period: POLARx FIT Substudy
Arm/Group | FROzEN
Started | 54 (Treatment = 50 Consent Ineligible = 1 Intent = 3)
Pre-Discharge | 50
3 Month Follow Up | 50
6 Month Follow Up | 50
12 Month Follow Up | 49
Completed | 49
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- FROzEN Non Roll-In Treatment Subjects; POLARx FIT Sub-study: Subjects undergoing cardiac ablation procedure with the Boston Scientific Cardiac Cryoablation System
  Boston Scientific Cardiac Cryoablation System: The Boston Scientific Cardiac Cryoablation System is intended for ablation and electrical mapping of the pulmonary veins for pulmonary vein isolation (PVI) in the ablation treatment of patients with paroxysmal atrial fibrillation (PAF).The main devices and components of the system consists of the following:
  * POLARx™ or POLARx FIT Cryoablation Catheter
  * POLARMAP™ Catheter
  * POLARSHEATH™
  * SMARTFREEZE™ Console
  * Diaphragm Movement Sensor (DMS)
  * Related Accessories
- Total: Total of all reporting groups
Arm/Group | FROzEN Non Roll-In Treatment Subjects | POLARx FIT Sub-study | Total
Number analyzed (Participants) | 325 | 50 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11) | 64 (13) | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 23 | 147
  Male | 201 | 27 | 228
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Native American | 1 | 0 | 1
  Asian | 35 | 0 | 35
  Black | 4 | 1 | 5
  Pacific Islander | 0 | 0 | 0
  White | 274 | 49 | 323
  Other | 1 | 0 | 1
  Race Undisclosed | 12 | 0 | 12
Height [Mean (Standard Deviation); unit: cm] | 174 (10) | 173 (10) | 174 (10)
Weight [Mean (Standard Deviation); unit: kg] | 86 (19) | 93 (22) | 87 (20)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29 (6) | 31 (7) | 29 (6)
Pulse [Mean (Standard Deviation); unit: bpm] | 67 (14) | 66 (13) | 67 (14)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 133 (18) | 134 (16) | 133 (18)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 79 (11) | 76 (9) | 79 (11)
CHA2DS2-VASc Score [Count of Participants; unit: Participants] — The CHA2DS2-VASc Score is a medical scale that refers to the various factors influencing the risk of stroke and other vascular incidents in patients with atrial fibrillations. A higher score indicates a higher risk.
  Participants
    0 | 63 | 3 | 66
    1 | 82 | 15 | 97
    2 | 92 | 16 | 108
    3 | 59 | 5 | 64
    4 | 21 | 6 | 27
    5 | 8 | 4 | 12
    6 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Primary Safety Events at 12 Months Post-procedure (Acute and Chronic Events) Using the Boston Scientific Cardiac Cryoablation System With POLARx Cryoablation Balloon Catheter Models
Description: This measure reports the observed safety event-free rate at 12 Months follow up for all Non Roll-In treatment and intent subjects. The safety events are a composite of procedure-related and device-related adverse events. 7 days (Death, Myocardial infarction, Transient ischemic attack, Stroke/ Cerebrovascular accident, Vascular access complications, Mitral or tricuspid valvular damage, Thromboembolism/ Air embolism leading to a life-threatening event such as a ventricular arrhythmia, stroke, pulmonary embolism, or myocardial infarction and, thromboembolic events that result in permanent injury, require intervention for treatment or prolongs or require hospitalization for more than 48 hours, Gastroparesis/injury to vagus nerve, Pneumothorax, Pulmonary edema/heart failure AV block); 30 days (Cardiac tamponade/perforation); 12 months: (Atrial esophageal fistula, Severe Pulmonary vein stenosis, Persistent phrenic nerve palsy .
Time Frame: 12 Months
Population: Non Roll-In Treatment and intent Subjects
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- FROzEN Non Roll-In Subjects: Subjects undergoing cardiac ablation procedure with the Boston Scientific Cardiac Cryoablation System
  Boston Scientific Cardiac Cryoablation System: The Boston Scientific Cardiac Cryoablation System is intended for ablation and electrical mapping of the pulmonary veins for pulmonary vein isolation (PVI) in the ablation treatment of patients with paroxysmal atrial fibrillation (PAF).The main devices and components of the system consists of the following:
  * POLARx™ or POLARx FIT Cryoablation Catheter
  * POLARMAP™ Catheter
  * POLARSHEATH™
  * SMARTFREEZE™ Console
  * Diaphragm Movement Sensor (DMS)
  * Related Accessories
Arm/Group | FROzEN Non Roll-In Subjects
Number analyzed (Participants) | 326
Percentage of participants | 96 [93.8 to NA] — One sided confidence interval

2. Primary Outcome: Percentage of Participants With Freedom From Treatment Failure at 12 Months Post-procedure Using the Boston Scientific Cardiac Cryoablation System With POLARx Cryoablation Balloon Catheter Models
Description: Freedom from the composite of: Failure to achieve acute procedural success in the index procedure or repeat procedure during the blanking period; Use of amiodarone post index procedure; Surgical treatment for AF/AFL/AT post index procedure; Use of non-study ablation catheter for AF targets in the index procedure or repeat procedure during the blanking period; More than one repeat procedure with the POLARx catheter during the blanking period (90 days post index procedure); Documented AF, or new onset of AF or AT event 91-365 days post index procedure; Any of the following for AF, or new onset of AF or AT 91-365 days post index procedure: Repeat procedure - Electrical and/or pharmacological cardioversion for AF/AFL/AT - Prescribed AAD consisting of any Class I/III, including Amiodarone, and any Class II/IV medications taken for control of AF, AT, AFL recurrence
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FROzEN Non Roll-In Subjects
Number analyzed (Participants) | 325
Percentage of participants | 59.9 [55.2 to NA] — One sided confidence interval

3. Primary Outcome: Percentage of Participants With Freedom From Primary Safety Events at 3 Months Post Procedure Using the Boston Scientific Cardiac Cryoablation System With POLARx FIT Cryoablation Balloon Catheter Models
Description: Composite of procedure-related and device-related adverse events. 7 days post index procedure or hospital discharge, whichever is later, unless denoted as events counting through 3 months post index procedure (Death, Myocardial infarction, Major Vagal Nerve Injury/Gastroparesis, Transient ischemic attack, Stroke/Cerebrovascular accident, Thromboembolism, Cardiac tamponade/perforation, Pneumothorax, Major vascular access complications, Pulmonary edema/heart failure, AV block, Atrial esophageal fistula, severe pulmonary vein stenosis (≥70% reduction in the diameter of the PV or PV branch from baseline), Persistent phrenic nerve palsy)
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | POLARx FIT Sub-Study
Number analyzed (Participants) | 50
Percentage of participants | 100 [92.9 to 100]

4. Primary Outcome: Percentage of Participants With Acute Procedural Success Defined as the Achievement of Electrical Isolation of All PVs by Using the Boston Scientific Cardiac Cryoablation System With POLARx Fit Cryoablation Balloon Catheter Models
Description: The primary effectiveness endpoint is the rate of acute procedural success where acute procedural success is defined as the achievement of electrical isolation of all PVs by using the Cardiac Cryoablation System with the POLARx FIT cryoablation balloon catheter models (with treatment applied at 28 mm or 31 mm balloon size per physician discretion). Electrical isolation of a PV is demonstrated by entrance and exit block.
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | POLARx FIT Sub-Study
Number analyzed (Participants) | 50
Percentage of participants | 100 [92.9 to 100]

5. Secondary Outcome: Percentage of Participants With Acute Procedural Success Defined as the Achievement of Electrical Isolation of All PVs by Using the Boston Scientific Cardiac Cryoablation System With POLARx Cryoablation Balloon Catheter
Description: The achievement of electrical isolation of all PVs by using the POLARx Cardiac Cryoablation System. Electrical isolation of a PV is demonstrated by entrance and exit block.
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FROzEN Non Roll-In Subjects
Number analyzed (Participants) | 325
Percentage of participants | 95.69 [92.88 to 97.63]

6. Secondary Outcome: Number of Participants With Freedom From Reportable Adverse Events at 12 Months Post Procedure Using the Boston Scientific Cardiac Cryoablation System With POLARx Cryoablation Balloon Catheter Models
Description: * All Serious Adverse Events
  * All Study Procedure-Related Adverse Events
  * All Study Device-Related Adverse Events
  * All Study Device Deficiencies
  * Unanticipated Adverse Device Effects/Unanticipated Serious Adverse Device Effects previously not defined in Investigator's Brochure or DFU
Time Frame: 12 months
Population: The total population represents all Non-Roll In (336) and Roll in (63) enrolled subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FROzEN
Number analyzed (Participants) | 399
Participants | 254

7. Secondary Outcome: Percentage of Participants With Freedom From Safety Events at 12 Months Post Procedure Using the Boston Scientific Cardiac Cryoablation System Using the Boston Scientific Cardiac Cryoablation System With POLARx FIT Cryoablation Balloon Catheter Models
Description: The following events will be counted through 7 days post index procedure or hospital discharge, whichever is later: Death, Myocardial infarction, Major Vagal Nerve Injury/Gastroparesis, Transient ischemic attack, Stroke/Cerebrovascular accident, Thromboembolism, Pneumothorax, Major vascular access complications, Pulmonary edema/heart failure, AV block. The following event will be counted through 30 days post index procedure: Cardiac tamponade/perforation. The following events will be counted through 12 months post index procedure: Atrial esophageal fistula, Severe pulmonary vein stenosis (≥70% reduction in the diameter of the PV or PV branch from baseline), Persistent phrenic nerve palsy.
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | POLARx FIT Sub-Study
Number analyzed (Participants) | 50
Percentage of participants | 100 [92.9 to NA] — One sided Confidence interval

8. Secondary Outcome: Percentage of Participants With Freedom From Treatment Failure at 12 Months Post-procedure Using the Boston Scientific Cardiac Cryoablation System With POLARx FIT Cryoablation Balloon Catheter Models
Description: Freedom from the composite of: Failure to achieve acute procedural success in the index procedure or repeat procedure during the blanking period; Use of amiodarone post index procedure; Surgical treatment for AF/AFL/AT post index procedure; Use of non-study ablation catheter for AF targets in the index procedure or repeat procedure during the blanking period; More than one repeat procedure with the Cryoablation System during the blanking period (90 days post index procedure); Documented AF, or new onset of AF or AT event 91-365 days post index procedure; Any of the following for AF, or new onset of AF or AT 91-365 days post index procedure: Repeat procedure - Electrical and/or pharmacological cardioversion for AF/AFL/AT - Prescribed AAD consisting of any Class I/III, including Amiodarone, and any Class II/IV medications taken for control of AF, AT, AFL recurrence
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | POLARx FIT Sub-Study
Number analyzed (Participants) | 50
Percentage of participants | 78 [66.5 to NA] — One-sided Confidence Interval

9. Other Pre Specified Outcome: Percentage of Participants With Freedom From Recurrence
Description: The following analysis looks at the recurrence free rate of individual atrial arrhythmia types as documented on a rhythm monitoring device post- blanking period.
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FROzEN Non Roll-In Subjects
Number analyzed (Participants) | 325
Percentage of participants | 79.9 [75.9 to NA] — One sided confidence interval

10. Post Hoc Outcome: Percentage of Participants With Freedom From Treatment Failure With Updated AAD Definition at 12 Months Post-procedure Using the Boston Scientific Cardiac Cryoablation System With POLARx Cryoablation Balloon Catheter Models
Description: In this sensitivity analysis, subjects were counted as primary effectiveness failures only if they were taking a new AAD not prescribed prior to index procedure or a higher dose of an AAD than they were previously prescribed.
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FROzEN Non Roll-In Subjects
Number analyzed (Participants) | 325
Percentage of participants | 71.6 [67.2 to NA] — One sided confidence interval

ADVERSE EVENTS:
Time Frame: Through 12 Months
Groups:
- FROzEN Non Roll In Treatment and Attempt Subjects; FROzEN Roll In Treatment Subjects; POLARx FIT Treatment Subjects: Subjects undergoing cardiac ablation procedure with the Boston Scientific Cardiac Cryoablation System
  Boston Scientific Cardiac Cryoablation System: The Boston Scientific Cardiac Cryoablation System is intended for ablation and electrical mapping of the pulmonary veins for pulmonary vein isolation (PVI) in the ablation treatment of patients with paroxysmal atrial fibrillation (PAF).The main devices and components of the system consists of the following:
  * POLARx™ or POLARx FIT Cryoablation Catheter
  * POLARMAP™ Catheter
  * POLARSHEATH™
  * SMARTFREEZE™ Console
  * Diaphragm Movement Sensor (DMS)
  * Related Accessories
Arm/Group | FROzEN Non Roll In Treatment and Attempt Subjects | FROzEN Roll In Treatment Subjects | POLARx FIT Treatment Subjects
All-Cause Mortality (participants affected / at risk) | 1/336 | 1/60 | 0/50
Serious Adverse Events (participants affected / at risk) | 33/326 | 10/60 | 4/50
Other Adverse Events (participants affected / at risk) | 86/326 | 16/60 | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FROzEN Non Roll In Treatment and Attempt Subjects (N=326) | FROzEN Roll In Treatment Subjects (N=60) | POLARx FIT Treatment Subjects (N=50)
Angina/ chest pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0)
Edema (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 6 (6) | 0 (0) | 1 (1)
Chest pain-other (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Fever and/or virus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 3 (5) | 2 (2) | 1 (1)
Integumentary (General disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Atrial Tachycardia/ Other SVT (e.g. AVRT, AVNRT, EAT) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple Symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Abnormal lab values (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cancer (General disorders) | 1 (1) | 2 (2) | 0 (0)
Hematological (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0)
Physical Trauma (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary (General disorders) | 0 (0) | 1 (2) | 0 (0)
1st Degree AV block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atypical (Type II) Atrial Flutter (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertensive/ Hypertensive crisis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular Tachycardiac (VT)/ Monomorphic VT (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
COPD Exacerbation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Genitourinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Neurological (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Vasovagal Reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FROzEN Non Roll In Treatment and Attempt Subjects (N=326) | FROzEN Roll In Treatment Subjects (N=60) | POLARx FIT Treatment Subjects (N=50)
Procedure related Pulmonary (including cough, hemoptysis) (Surgical and medical procedures) | 5 (5) | 0 (0) | 0 (0)
Atrial (Type I) Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 5 (5) | 6 (6) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain- other (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Conduction pathway injury (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Hypertension/ Hypertensive crisis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension/ Orthostatic hypotension (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Multiple symptoms (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular Tachycardia (VT)/ Monomorphic VT (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Fever and/or virus (General disorders) | 1 (1) | 2 (2) | 2 (2)
Head, Eyes, Ears, Nose, Throat (HEENT) (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hematological (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Neurological (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Physical Trauma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary (General disorders) | 1 (1) | 0 (0) | 0 (0)
Renal (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Procedure related Anesthesia/ sedation (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0)
Atrial tachycardia/ Other SVT (e.g AVRT, AVNRT, EAT) (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Localized infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Psychological (General disorders) | 0 (0) | 1 (1) | 0 (0)
Premature atrial contractions (PAC) (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ablation induced Arrhythmia (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0)
Angina/ chest pain (Surgical and medical procedures) | 5 (5) | 0 (0) | 0 (0)
Atrial Flutter (not specified) (Surgical and medical procedures) | 6 (6) | 0 (0) | 0 (0)
Bleeding related to anticogulation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Edema (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Embolism - air (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Gasteroparesis (Surgical and medical procedures) | 5 (5) | 1 (1) | 0 (0)
Hematoma (Surgical and medical procedures) | 13 (13) | 0 (0) | 0 (0)
Myocardial Infarction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Myocardial Perforation with tamponade (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Oozing/ bleeding (Surgical and medical procedures) | 7 (7) | 0 (0) | 0 (0)
Pain (non-cardiovascular) (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Surgical and medical procedures) | 13 (13) | 1 (1) | 0 (0)
Phrenic Nerve Injury temporary (Surgical and medical procedures) | 10 (10) | 3 (3) | 0 (0)
Pleuritis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Post procedure infection/ Sepsis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Post procedure wound discomfort (Surgical and medical procedures) | 5 (5) | 2 (2) | 0 (0)
Procedure related allergic reactions/ adverse drug reaction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Procedure related anesthesia/ sedation (Surgical and medical procedures) | 2 (2) | 1 (3) | 0 (0)
Procedure related gastrointestinal (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Procedure related hypertension (Surgical and medical procedures) | 3 (3) | 0 (0) | 0 (0)
Procedure related Neurological (non-TIA, non-stroke, dysphagia, speech disturbance/ dysarthria) (Surgical and medical procedures) | 4 (4) | 0 (0) | 0 (0)
Pulmonary Edema (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Right atrial (type 1) atrial flutter (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall have the right to publish the Results, provided that before publishing, Institution and Investigator shall submit copies of any proposed publication or presentation to Sponsor for review at least sixty (60) days in advance of submission for publication or presentation to a publisher or other third party. In addition, Sponsor may extend such review period for another ninety (90) days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04133168/Prot_SAP_000.pdf